CLINICAL TRIAL: NCT02257021
Title: Study of Pharmacokinetic Interaction Between Tipranavir and BILR 355 BS Plus Ritonavir
Brief Title: Pharmacokinetic Interaction Between Tipranavir and BILR 355 BS Plus Ritonavir in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1188.7
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir

ARMS (2):
- Tipranavir and high dose of ritonavir plus BILR 355 BS (Experimental)
  Interventions: Drug: BILR 355 BS; Drug: Tipranavir; Drug: High dose of ritonavir
- BILR 355 BS with low dose of ritonavir (Experimental)
  Interventions: Drug: BILR 355 BS; Drug: Low dose of ritonavir

INTERVENTIONS:
Drug: BILR 355 BS
Drug: Tipranavir
  Arms: Tipranavir and high dose of ritonavir plus BILR 355 BS
Drug: Low dose of ritonavir
  Arms: BILR 355 BS with low dose of ritonavir
Drug: High dose of ritonavir
  Arms: Tipranavir and high dose of ritonavir plus BILR 355 BS

SUMMARY:
To determine the effect of BILR 355/r on tipranavir/r pharmacokinetics and the effect of tipranavir/r on BILR 355 BS pharmacokinetics

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19 and <60 years
* BMI ≥18.5 and BMI ≤29.9 kg/m2
* Ability to give signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and the local regulations

Exclusion Criteria:

* Current (symptomatic within the last 30 days) and medically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Currently active (symptomatic within the last 30 days) diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 hours) within one month prior to administration of study drug or during the trial (review with clinical monitor if questionable)
* Use of drugs within 10 days prior to administration or during the trial, which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation (review with clinical monitor if questionable)
* Participation in another trial with an investigational drug within one month prior to administration or during the trial
* Current smoker or smoked within the past 30 days
* Alcohol (more than 60 g/day) or drug abuse (positive urine test for illicit prescription or non-prescription drugs or drugs of abuse)
* Recent blood donation (more than 100 mL within 56 days prior to administration or during the trial)
* Excessive physical activities (within 1 week prior to study drug administration or during the trial)
* Any laboratory value outside the normal reference range that is of clinical relevance at screening, according to the judgment of the investigator
* Inability to comply with dietary regimen required by the protocol
* Chronic or relevant acute infections
* Infected with hepatitis B or hepatitis C viruses (defined as either being hepatitis B surface antigen, or hepatitis C antibody positive)
* HIV-1 infected as defined by a positive HIV ELISA test

Ages: 19 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2005-02; Primary Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of tipranavir and BILR 355 BS in plasma over one dosing interval (12 hours) at steady state (AUC0-12h,ss) | up to 18 days after start of treatment
Maximum measured concentration of tipranavir and BILR 355 BS in plasma at steady state over a dosing interval τ (Cmax,ss) | up to 18 days after start of treatment

SECONDARY OUTCOMES:
Apparent clearance of BILR 355 BS, tipranavir and ritonavir in plasma following extravascular administration at steady state (CL/F,ss) | up to 18 days after start of treatment
Time from dosing to the maximum concentration of BILR 355 BS, tipranavir and ritonavir in plasma at steady state (tmax,ss) | up to 18 days after start of treatment
Terminal half-life of BILR 355 BS, tipranavir and ritonavir in plasma at steady state (t1/2,ss) | up to 18 days after start of treatment
Apparent volume of distribution of BILR 355 BS, tipranavir and ritonavir during the terminal phase λz at steady state following an extravascular dose (Vz/F,ss) | up to 18 days after start of treatment
Area under the concentration-time curve of ritonavir in plasma over one dosing interval (12 hours), (AUC0-12h) | up to 18 days after start of treatment
Maximum measured concentration of ritonavir in plasma at steady state over a dosing interval τ (Cmax,ss) | up to 18 days after start of treatment
Measured concentration of BILR 355 BS, tipranavir and ritonavir in plasma 12 hours post last dose at steady state (Cp12h,ss) | up to 18 days after start of treatment
Number of participants with clinically relevant changes in laboratory parameters | up to 28 days after start of treatment
Number of participants with clinically relevant changes in vital signs (blood pressure, pulse rate) | up to 28 days after start of treatment
Number of participants with clinically relevant changes in 12-lead ECG | up to 14 days after start of treatment
Number of participants with adverse events | Up to 7 weeks